CLINICAL TRIAL: NCT05237414
Title: Forgetting Alcohol: a Double-blind, Randomized Controlled Trial Investigating Memory Inhibition Training in Young Binge Drinkers.
Brief Title: Combining Cognitive Training With tDCS to Enhance Memory Inhibition in Young Binge Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Eduardo López-Caneda, Postdoctoral Researcher, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PTDC/PSI-ESP/28672/2017; CE.CSH 078/2018 (Other: Ethics Committee of University of Minho); PTDC/PSI-ESP/28672/2017 (Other Grant/Funding Number: Portuguese Foundation for Science and Technology)
Record Dates: First submitted 2022-01-17; First posted 2022-02-14 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Binge Drinking
Keywords: Alcohol; Craving; Binge Drinking; College Students; Memory Inhibition; Alcohol-Related Memories; Randomized Controlled Trial; Intervention Protocol; Cognitive Training; Transcranial Direct-Current Stimulation (tDCS); Electroencephalography (EEG); Event-Related Potentials (ERPs); Functional Connectivity
MeSH Terms: conditions — Binge Drinking | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: BDs will be randomly distributed for one of three training conditions: Combined Training (i.e, active tDCS and active CT), Cognitive Training (i.e., sham tDCS and active CT), and Control (i.e., sham tDCS and sham CT).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Binge Drinkers with Combined Intervention (active CT + active tDCS) (Experimental): Subjects will perform a variation of the TNTA task (Anderson & Green, 2001; López-Caneda et al., 2019) to enhance the suppression of alcohol-related memories. The Learning phase will be composed of 2 blocks of 12-image pairs (as there is no a baseline block), and in the TNT phase, all the stimuli to be inhibited will be alcohol-related images. After the Learning Phase, active neuromodulation will be performed using tDCS. Twenty minutes of 2 mA direct current will be applied on the scalp using a saline-soaked pair of 35 cm2 surface sponge electrodes, through an Eldith DC Stimulator Plus (Neuroconn, Germany). To stimulate the right DLPFC, the anodal electrode will be placed over F4 according to the 10-20 international system for EEG electrode placement. The cathode electrode will be over the contralateral supraorbital area. The current fade in for 15 seconds, is constant at 2 mA for 20 minutes, and then fade out for 15 seconds.
  Interventions: Device: Active tDCS; Behavioral: Active CT
- Binge Drinkers with Cognitive Intervention (active CT + sham tDCS) (Experimental): Subjects perform the variation of the TNTA task for active CT. After the Learning Phase, sham neuromodulation is performed using the same montage of the active tDCS. However, the electric current fade in during 15 seconds until reaching 2 mA, then is constant at 2 mA for 15 seconds and fade out for 15 seconds. There is no current for the rest of the time.
  Interventions: Device: Sham tDCS; Behavioral: Active CT
- Binge Drinkers with Control Intervention (sham CT + sham tDCS) (Sham Comparator): Subjects will perform a variation of the TNTA task, where the Learning phase also have only two blocks of 12-image pairs. However, in this case the TNT phase is replaced by a Forced-Choice Reaction Time (FCRT) task, during which the participants only must categorize alcoholic and non-alcoholic images answering to the question "What type of beverage was there in the image?" (answer: "Alcoholic drink" or "Non-alcoholic drink"); thus, they do not have to inhibit the memories related to the alcoholic images. During this phase, sham neuromodulation will be performed using the same montage of the active tDCS. The electric current fade in during 15 seconds until reaching 2 mA, then is constant at 2 mA for 15 seconds and fade out for 15 seconds, while a sham memory inhibition CT is performed.
  Interventions: Device: Sham tDCS; Behavioral: Sham CT
- Non/Low-Drinkers (No Intervention): No intervention.

INTERVENTIONS:
Device: Active tDCS — 20 minutes of 2.0 mA direct current applied over the right DLPFC
  Arms: Binge Drinkers with Combined Intervention (active CT + active tDCS)
Device: Sham tDCS — 15 seconds of 2.0 mA direct current applied over the right DLPFC
  Arms: Binge Drinkers with Cognitive Intervention (active CT + sham tDCS); Binge Drinkers with Control Intervention (sham CT + sham tDCS)
Behavioral: Active CT — Active memory inhibition CT (i.e., training of memory inhibition specifically for alcohol-related memories).
  Arms: Binge Drinkers with Cognitive Intervention (active CT + sham tDCS); Binge Drinkers with Combined Intervention (active CT + active tDCS)
Behavioral: Sham CT — Sham memory inhibition CT (i.e., participants have to categorize alcoholic and non-alcoholic images but they do not have to inhibit the memories related to these images).
  Arms: Binge Drinkers with Control Intervention (sham CT + sham tDCS)

SUMMARY:
This study protocol aims to examine the behavioral and electroencephalographic (EEG) correlates of memory inhibition (MI) among college binge drinkers (BDs). A second objective is to evaluate an alcohol-specific MI training protocol using cognitive training (CT) and transcranial direct current stimulation (tDCS) while its effects on behavioral and EEG outcomes are assessed. Along with poor MI abilities, we hypothesized that BDs would show alterations in the amplitude of several event-related potentials (ERPs) linked to MI (e.g., N2 and late parietal positivity) as well as abnormal functional connectivity (FC) patterns within/between regions associated with MI (e.g., dorsolateral prefrontal cortex [DLPFC] and hippocampal/parahippocampal regions). Results should also demonstrate the effectiveness of the training protocol, with BDs exhibiting an improved capacity to suppress alcohol-related memories after both combined and cognitive MI training, along with a significant reduction in alcohol use and craving in the short/medium-term. Furthermore, this protocol should also lead to significant modifications in the ERP and FC patterns, reflecting stronger MI capabilities and reduced alcohol cue reactivity in trained BD participants.

DETAILED DESCRIPTION:
The present study protocol aims to examine the behavioral and EEG correlates of MI, specifically those related to the suppression of alcohol-related memories, among young BDs. For this purpose, 45 BDs and 45 age-matched non/low-drinkers (N/LDs) will be assessed by EEG while performing the Think/No-Think Alcohol (TNTA) task, a paradigm that evaluates alcohol-related MI (Pre-training EEG assessment). The TNTA is divided into three phases: 1) the Learning phase, 2) the Think/No-Think (TNT) phase and 3) the Memory-Test phase. During the learning phase, participants will be asked to associate and memorize 36 pairs of neutral objects + alcoholic/non-alcoholic pictures. Then, only the neutral objects will be presented, and participants will have to try to remember the picture (alcoholic/non-alcoholic image) that was associated with this neutral object and answer three questions about the beverage depicted, the orientation of the picture and the number of people present in it. After the learning phase, the Think/No -Think phase will comprehend two conditions: in the Think condition (depicted in the neutral images with a green frame),participants are presented with the object and they will be instructed to "think of the previously learned alcoholic/non-alcoholic picture and keep it in mind during the entire presentation of the object". In the No-Think condition (depicted by neutral images with a red frame) they will be asked "not to let the previously associated picture enter your consciousness". In the memory test phase, the 36 neutral images will be presented again, including the 12 neutral objects of the baseline condition that were not presented in the TNT phase. Participants will be asked to recall - answering the same three questions of the learning phase - the image (alcoholic/non-alcoholic) that was initially associated with the neutral object.

During this pre-training session, psychological (i.e., craving levels), behavioral (i.e., alcohol consumption, recall accuracy and MI performance), and neurofunctional (i.e., ERPs and FC) variables will be assessed.

In addition, this study aims to evaluate an alcohol-specific MI intervention protocol using cognitive training and tDCS while its effects on behavioral and EEG outcomes are assessed. For that, BDs will be randomly assigned to one of three training groups: combined intervention (active CT and active tDCS applied over the right DLPFC), cognitive intervention (active CT and sham tDCS), or control intervention (sham CT and sham tDCS). Training will occur in three consecutive days (i.e., Tuesday, Wednesday, and Thursday), in three sessions. MI will be re-assessed in BDs after the last training session through a post-training EEG assessment. N/LDs will only perform the pre-training EEG assessment. Alcohol use and craving will also be measured both 10-days and 3-months post-training in order to monitor short- and medium-term effects of the MI training in the alcohol craving and consumption levels. Furthermore, behavioral and EEG data will be collected during the performance of an alcohol cue reactivity (ACR) task before and after the MI training sessions, in order to evaluate potential attentional bias towards alcoholic stimuli. Overall, this intervention protocol aims to investigate whether this training is able 1) to enhance MI capabilities and to reduce alcohol attentional bias, and 2) to decrease craving and/or alcohol use -monitoring up to three months after protocol implementation- in trained BD participants.

ELIGIBILITY:
Inclusion Criteria:

* College students
* Age 18-24 years
* Binge Drinkers: report (i) drinking 5 or more drinks on one occasion at least once a month, and (ii) drinking at a speed of at least two drinks per hour during these episodes (which brings blood alcohol concentration to 0.08 gram percent or above).
* Non/Low-Drinkers: report (i) never drinking 5 or more drinks on one occasion and (ii) having an AUDIT score ≤ 4.

Exclusion Criteria:

* Use of illegal drugs except cannabis (as determined by the Drug Use Disorders Identification Test-Extended [DUDIT-E; Berman, Bergman, Palmstierna & Schlyter, 2007);
* Alcohol abuse (i.e., AUDIT ≥ 20);
* Consumption of medical drugs with psychoactive effects (e.g., sedatives or anxiolytics) during the two weeks before the experiment;
* Personal history of psychopathological disorders (according to DSM-V criteria);
* History of traumatic brain injury or neurological disorder;
* Family history of alcoholism or diagnosis of other substance abuse;
* Occurrence of one or more episodes of loss of consciousness for more than 20 minutes;
* Non-corrected sensory deficits;
* Global Severity Index (GSI) > 90 (Symptom Checklist-90-Revised questionnaire [SCL-90-R]; Derogatis, 1983) or a score above 90 in at least two of the symptomatic dimensions.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Behavioral Memory Inhibition Performance | At baseline (pre-training)
  MI, specifically alcohol-related MI, will be assessed using the TNTA task. Percentage of correct responses (for Think, No-Think and Baseline items) in the TNTA task will be computed according to the following formula: ((number of correctly recalled items)/(number of previously learned items))×100. Correct responses correspond to the items learned during the learning phase and correctly recalled during the memory test phase.
Behavioral Memory Inhibition Performance | 1day after MI training
  MI, specifically alcohol-related MI, will be assessed using the TNTA task. Percentage of correct responses (for Think, No-Think and Baseline items) in the TNTA task will be computed according to the following formula: ((number of correctly recalled items)/(number of previously learned items))×100. Correct responses correspond to the items learned during the learning phase and correctly recalled during the memory test phase.
EEG correlates of Memory Inhibition Performance - N2 ERP component | At baseline (pre-training)
  After EEG data collection, the mean amplitude of N2 component will be analyzed.
EEG correlates of Memory Inhibition Performance - N2 ERP component | 1day after MI training
  After EEG data collection, the mean amplitude of N2 component will be analyzed.
EEG correlates of Memory Inhibition Performance - LPP ERP component | At baseline (pre-training)
  After EEG data collection, the mean amplitude of Late Parietal Positivity (LPP) will be analyzed.
EEG correlates of Memory Inhibition Performance - LPP ERP component | 1day after MI training
  After EEG data collection, the mean amplitude of Late Parietal Positivity (LPP) will be analyzed.
EEG correlates of Memory Inhibition Performance - Frontal slow wave (FSW) ERP component | At baseline (pre-training)
  After EEG data collection, the mean amplitudes of FSW will be analyzed
EEG correlates of Memory Inhibition Performance - Frontal slow wave (FSW) ERP component | 1day after MI training
  After EEG data collection, the mean amplitudes of FSW will be analyzed
EEG correlates of Memory Inhibition Performance - Functional connectivity (FC) | At baseline (pre-training)
  FC patterns within/between regions associated with MI (e.g., DLPFC and hippocampal/parahippocampal regions) will also be assessed.
EEG correlates of Memory Inhibition Performance - Functional connectivity (FC) | 1day after MI training
  FC patterns within/between regions associated with MI (e.g., DLPFC and hippocampal/parahippocampal regions) will also be assessed.
Alcohol Cue Reactivity - Emotional measures | At baseline (pre-training)
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set (Pronk, van Deursen, Beraha, Larsen & Wiers, 2015).
  The emotional responses for each image in terms of valence and arousal task, will be registered using the Self-Assessment Manikin (valence: from 1 = "very unpleasant" to 9 ="very pleasant"; arousal: from 1 = "not arousing" to 9 = "highly arousing") during the ACR task.
Alcohol Cue Reactivity - Emotional measures | 1day after MI training
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set (Pronk, van Deursen, Beraha, Larsen & Wiers, 2015).
  The emotional responses for each image in terms of valence and arousal task, will be registered using the Self-Assessment Manikin (valence: from 1 = "very unpleasant" to 9 ="very pleasant"; arousal: from 1 = "not arousing" to 9 = "highly arousing") during the ACR task.
EEG correlates of Alcohol Cue Reactivity - P1 ERP component | At baseline (pre-training)
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set. After EEG data collection, the mean amplitude of the P1 for alcoholic and non-alcoholic images of ACR task will be analyzed.
EEG correlates of Alcohol Cue Reactivity - P1 ERP component | 1day after MI training
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set. After EEG data collection, the mean amplitude of the P1 for alcoholic and non-alcoholic images of ACR task will be analyzed.
EEG correlates of Alcohol Cue Reactivity - N1 ERP component | Baseline (pre-training)
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set. After EEG data collection, the mean amplitude of the N1 for alcoholic and non-alcoholic images of ACR task will be analyzed.
EEG correlates of Alcohol Cue Reactivity - N1 ERP component | 1day after MI training
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set. After EEG data collection, the mean amplitude of the N1 for alcoholic and non-alcoholic images of ACR task will be analyzed.
EEG correlates of Alcohol Cue Reactivity - P2 ERP component | Baseline (pre-training)
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set. After EEG data collection, the mean amplitude of the P2 for alcoholic and non-alcoholic images of ACR task will be analyzed.
EEG correlates of Alcohol Cue Reactivity - P2 ERP component | 1day after MI training
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set. After EEG data collection, the mean amplitude of the P2 for alcoholic and non-alcoholic images of ACR task will be analyzed.
EEG correlates of Alcohol Cue Reactivity - Functional Connectivity | Baseline (pre-training)
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set. After EEG data collection, FC patterns of visual and attentional networks will be assessed.
EEG correlates of Alcohol Cue Reactivity - Functional Connectivity | 1day after MI training
  The reactivity to alcoholic cues will be assessed using the ACR task. The full task includes a total of 80 trials with 40 alcoholic and 40 non-alcoholic images obtained from the Amsterdam Beverage Picture Set. After EEG data collection, the FC patterns of visual and attentional networks will be assessed.
Alcohol Consumption - Drinking pattern | Screening Visit (Clinical Interview)
  The Alcohol Use Disorder Identification Test (AUDIT; Babor, Higgins-Biddle, Saunders, Monteiro, 2001) will be administered to characterize the drinking pattern of the participants. AUDIT scores < 8 reveal low risk of alcohol use; scores between 8 and 15 represent a risky consumption; scores from 16 to 19 are considered a harmful intake pattern; and scores ≥ 20 indicate very high risk for alcohol dependence and warrant further diagnostic evaluation for alcohol dependence.
Alcohol Consumption - Drinking pattern | At baseline (pre-training)
  The Alcohol Use Disorder Identification Test (AUDIT; Babor, Higgins-Biddle, Saunders, Monteiro, 2001) will be administered to characterize the drinking pattern of the participants. AUDIT scores < 8 reveal low risk of alcohol use; scores between 8 and 15 represent a risky consumption; scores from 16 to 19 are considered a harmful intake pattern; and scores ≥ 20 indicate very high risk for alcohol dependence and warrant further diagnostic evaluation for alcohol dependence.
Alcohol Consumption - Drinking pattern | 10 days after MI training
  The Alcohol Use Disorder Identification Test (AUDIT; Babor, Higgins-Biddle, Saunders, Monteiro, 2001) will be administered to characterize the drinking pattern of the participants. AUDIT scores < 8 reveal low risk of alcohol use; scores between 8 and 15 represent a risky consumption; scores from 16 to 19 are considered a harmful intake pattern; and scores ≥ 20 indicate very high risk for alcohol dependence and warrant further diagnostic evaluation for alcohol dependence.
Alcohol Consumption - Drinking pattern | 3 months after MI training
  The Alcohol Use Disorder Identification Test (AUDIT; Babor, Higgins-Biddle, Saunders, Monteiro, 2001) will be administered to characterize the drinking pattern of the participants. AUDIT scores < 8 reveal low risk of alcohol use; scores between 8 and 15 represent a risky consumption; scores from 16 to 19 are considered a harmful intake pattern; and scores ≥ 20 indicate very high risk for alcohol dependence and warrant further diagnostic evaluation for alcohol dependence.
Alcohol consumption - Previous week | At baseline (pre-training)
  The number of drinks in the previous week will be assessed using the Alcohol Timeline Followback (TLFB)
Alcohol consumption - Previous week | 10-days after MI training
  The number of drinks in the previous week will be assessed using the Alcohol Timeline Followback (TLFB)
Alcohol consumption - Previous week | 3-months after MI training
  The number of drinks in the previous week will be assessed using the Alcohol Timeline Followback (TLFB)
Alcohol consumption - Typical weeks | Baseline (pre-training)
  The number of drinks during a standard/typical week and the frequency of typical weeks during the previous three months will be assessed using Typical and Atypical Drinking Diary (TADD).
Alcohol consumption - Typical weeks | 3-months after MI training
  The number of drinks during a standard/typical week and the frequency of typical weeks during the previous three months will be assessed using Typical and Atypical Drinking Diary (TADD).
Alcohol consumption - Atypical weeks | Baseline (pre-training)
  the number of drinks during an atypical week (i.e., week with a greater consumption of alcohol) and the frequency of atypical weeks during the previous three months will be assessed using Typical and Atypical Drinking Diary (TADD).
Alcohol consumption - Atypical weeks | 3-months after MI training
  the number of drinks during an atypical week (i.e., week with a greater consumption of alcohol) and the frequency of atypical weeks during the previous three months will be assessed using Typical and Atypical Drinking Diary (TADD).
Alcohol Craving - Short-term acute craving | Baseline (pre-training)
  Short-term alcohol craving levels will be assessed using the Alcohol Craving Questionnaire - Short form Revised (ACQ-SF-R) Portuguese version (Rodrigues et al., 2021). Total minimum score: 1 (low level of alcohol craving); Total maximum score: 7 (high level of alcohol craving)
Alcohol Craving - Short-term acute craving | 10-days after MI training
  Short-term alcohol craving levels will be assessed using the Alcohol Craving Questionnaire - Short form Revised (ACQ-SF-R) Portuguese version (Rodrigues et al., 2021). Total minimum score: 1 (low level of alcohol craving); Total maximum score: 7 (high level of alcohol craving)
Alcohol Craving - Short-term acute craving | 3-months after MI training
  Short-term alcohol craving levels will be assessed using the Alcohol Craving Questionnaire - Short form Revised (ACQ-SF-R) Portuguese version (Rodrigues et al., 2021). Total minimum score: 1 (low level of alcohol craving); Total maximum score: 7 (high level of alcohol craving)
Alcohol Craving - Past level of craving | Baseline (pre-training)
  alcohol craving levels during the past week will be evaluated using Penn Alcohol Craving Scale (PACS) Portuguese version (Pombo, Ismail & Cardoso, 2008). Total minimum score: 0 (low level of alcohol craving); Total maximum score: 36 (high level of alcohol craving)
Alcohol Craving - Past level of craving | 10-days after MI training
  alcohol craving levels during the past week will be evaluated using Penn Alcohol Craving Scale (PACS) Portuguese version (Pombo, Ismail & Cardoso, 2008). Total minimum score: 0 (low level of alcohol craving); Total maximum score: 36 (high level of alcohol craving)
Alcohol Craving - Past level of craving | 3-months after MI training
  alcohol craving levels during the past week will be evaluated using Penn Alcohol Craving Scale (PACS) Portuguese version (Pombo, Ismail & Cardoso, 2008). Total minimum score: 0 (low level of alcohol craving); Total maximum score: 36 (high level of alcohol craving)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo G. López-Caneda, PhD, Principal Investigator — University of Minho
Locations (1):
- School of Psychology, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez-Caneda E, Crego A, Campos AD, Gonzalez-Villar A, Sampaio A. The Think/No-Think Alcohol Task: A New Paradigm for Assessing Memory Suppression in Alcohol-Related Contexts. Alcohol Clin Exp Res. 2019 Jan;43(1):36-47. doi: 10.1111/acer.13916. Epub 2018 Nov 25. PMID 30375668
- [Derived] Almeida-Antunes N, Anton-Toro L, Crego A, Rodrigues R, Sampaio A, Lopez-Caneda E. Trying to forget alcohol: Brain mechanisms underlying memory suppression in young binge drinkers. Prog Neuropsychopharmacol Biol Psychiatry. 2024 Aug 30;134:111053. doi: 10.1016/j.pnpbp.2024.111053. Epub 2024 Jun 11. PMID 38871018
- [Derived] Almeida-Antunes N, Vasconcelos M, Crego A, Rodrigues R, Sampaio A, Lopez-Caneda E. Forgetting Alcohol: A Double-Blind, Randomized Controlled Trial Investigating Memory Inhibition Training in Young Binge Drinkers. Front Neurosci. 2022 Jun 29;16:914213. doi: 10.3389/fnins.2022.914213. eCollection 2022. PMID 35844233

DOCUMENTS (3):
  • Study Protocol (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT05237414/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT05237414/SAP_001.pdf
  • Informed Consent Form (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT05237414/ICF_002.pdf